CLINICAL TRIAL: NCT06396520
Title: Neuroimaging of Babies During Natural Sleep to Assess Typical Development and Cerebral Palsy
Acronym: NIBS-CP
Status: Recruiting | Type: Observational
Sponsor: Danish Research Centre for Magnetic Resonance (Other)
Collaborators: Hvidovre University Hospital (Other); Department of Pediatrics and Adolescent Medicine, Rigshospitalet, Denmark (Unknown)
Responsible Party: Sponsor
Other Study IDs: NIBS-CP
Record Dates: First submitted 2024-04-29; First posted 2024-05-02 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Cerebral Palsy; Infant Development; Development, Infant
Keywords: MRI; Brain development; Diffusion MRI; Motor development; Cognitive development; Normative modelling; Hand assessment for infants; Alberta Infant Motor scale; Motor functioning; Cerebral Palsy; Typically developing; Infants; Toddlers; Children; Peabody Developmental Motor Scales; Corticospinal tract; Motor system
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Typically developing infants: Born after gestational week 37, Uneventful birth, No known history of brain injury, No known neurological disorders
  Interventions: Other: No intervention, observational
- High Risk for Cerebral Palsy: Recruitment through CP-EDIT (Clinical trials.gov ID: NCT05835674), inclusion criteria.
  'Newborn-detectable risk-pathway'. Preterm birth with gestational age below 32 or birth weight below 1500 g and clinical concern, Moderate to severe brain injury (Papile grade 3 to 4 intraventricular haemorrhage, cystic periventricular leukomalacia, neonatal stroke, term hypoxic-ischaemic encephalopathy (≥35 weeks gestation at birth) or other significant neurological condition), History (e.g. neonatal seizures, Extra Corporal Membrane Oxygenation, meningitis, kernicterus, severe hypoglycemia) or neurological risk factors (brain malformation, increased tone), Parental concern and one of the factors above
  'Infant detectable risk-pathway'. Inability to sit independently by age 9 months, Hand function asymmetry or crawl asymmetry, Inability to take weight through the plantar surface of the feet, History (as above) or neurological risk factors, Parental concern and one of the factors above.
  Interventions: Other: No intervention, observational

INTERVENTIONS:
Other: No intervention, observational — No intervention, observational

SUMMARY:
Background: Early diagnosis of cerebral palsy (CP) is crucial, enabling intervention when neuroplasticity is at its highest. Magnetic resonance imaging (MRI) plays a vital role in CP diagnosis. Currently, diagnostic MRI of newborns and infants with suspected brain damage relies heavily on structural MR images. The current study aims to i) establish procedures for clinical infant and toddler MRI during natural sleep, ii) use advanced MRI sequences, such as advanced diffusion-weighted imaging (DWI), that may be more sensitive in detecting early brain damage, and iii) map relationships between early brain development, and motor function and development.

Methods: The NIBS-CP study will enroll approximately 200 infants either at risk for CP or typically developing. Infants will be followed longitudinally (for three waves) between 3 months and 2 years of age with cerebral MRI at 3 Tesla and comprehensive assessments of motor and cognitive functioning. The MRI protocol includes advanced diffusion-weighted imaging, high-resolution structural MRI, and MR spectroscopy. The motor and cognitive assessments include Hand Assessment in Infants, Alberta Infant Motor Scales, Hammersmith Infant Neurological Examination, Peabody Developmental Motor Scales, Bayley Scales of Infant Development, and Ages and Stages Questionnaires. NIBS-CP aims to establish normative material on early brain development of Danish children and conduct normative modeling of typical and atypical development to identify deviations in brain development at the level of the single child.

Discussion: Identifying predictive brain structural features of motor function and motor development is key to the future use of early MRI in the clinical work-up, as this promotes early diagnosis and (clinical) intervention strategies tailored to the individual child.

DETAILED DESCRIPTION:
Diagnostic magnetic resonance imaging (MRI) of newborns and infants with suspected brain damage is today based on conventional structural MR images with the focus on identifying major structural brain pathology. However, advanced MRI sequences, such as advanced diffusion-weighted imaging, may be more sensitive to detecting brain damage. The NeuroImaging of Babies during natural Sleep to assess typical development and CP (NIBS-CP) study is a longitudinal cohort study of infants and toddlers aged 3-24 months, aimed at studying early brain development in infants at risk of cerebral palsy (CP) and typically developing infants using advanced MRI sequences. The NIBS-CP cohort consists of:

1. Infants at risk for CP, recruited from the Cerebral Palsy: Early Diagnosis and Intervention Trial (CP-EDIT).

   The ongoing Danish CP-EDIT by principal investigator Professor Christina Høi-Hansen is registered with ClinicalTrials.gov ID NCT05835674. CP-EDIT will enroll 160 infants aged 3-11 months with CP or high risk of CP. Infants will be followed longitudinally with a large battery of motor, neurological, and cognitive assessments during the first two years of life. In addition, CP-EDIT contains information from patient journals on diagnostic MRI, but CP-EDIT does not include the collection of MRI scans as part of the study. For infants enrolled in CP-EDIT, participation in NIBS-CP only includes advanced MRI scans and parent-reported questionnaires. All neurological, motor, and cognitive assessments will be undertaken in CP-EDIT.
2. Typically developing infants, recruited specifically for NIBS-CP. For these infants, participation in NIBS-CP includes advanced MRI scans, neurological, motor, and cognitive assessments (similar to the ones included in CP-EDIT), and parent-reported questionnaires. NIBS-CP provides a control cohort of typically developing infants that will give rise to a normative Danish sample of early brain development to the infants at high risk of CP, as CP-EDIT does not include a control cohort of typically developing infants.

AIMS

The NIBS-CP project aims to:

1. Establish procedures for infant and toddler MRI during natural sleep without the use of sedation or GA at Hvidovre Hospital.
2. Employ advanced MRI sequences for scanning infants and toddlers, e.g., advanced diffusion-weighted imaging, high-resolution structural MRI, and MR spectroscopy, which are likely to be more sensitive in detecting brain injury and damage than conventional diagnostic MRI.
3. Initiate a cohort of typically developing infants and toddlers, and perform longitudinal advanced MRI of infants at high risk for CP. The NIBS-CP cohort will be used to:

   * Establish a dataset of normative material of early brain development of Danish children.
   * Conduct normative modeling of typical and atypical early brain development, i.e., analogous to growth charts, to inform about differences in brain development at the level of a single child.
   * Map relationships between early brain development, and motor function and development. Identifying predictive features of brain structure with MRI is key to the future use of early MRI in the clinical work-up, as these features may enable a better prediction of the prospects of motor function and motor development of the child.

HYPOTHESES

The primary hypotheses are that:

* Infants with CP will show reduced hand functioning which relates to decreased myelination and microstructural integrity primarily in the corticospinal tract.
* Infants with unilateral brain injuries will display asymmetrical hand functioning, which will be linked to asymmetrical corticospinal tract microstructure and myelination.

The secondary hypotheses are that:

* Reduced hand functioning and hand functioning asymmetry will also be related to:

  * decreased myelination and microstructural integrity in other key motor regions, such as the basal ganglia, motor cortex, cerebellum, and white matter tracts
  * the metabolic profile of the basal ganglia/internal capsule.
* Infants with CP will show reduced gross motor functioning, which relates to decreased myelination and microstructural integrity in key motor regions, such as the basal ganglia, motor cortex, cerebellum, and white matter tracts, e.g., the corticospinal tract.

Furthermore, the normative modeling framework, similar to pediatric growth curves, will be used to elucidate how individual infants with high risk for CP deviate from the norm on different brain outcome measures. The relationships between developing motor functioning and brain structural outcome measures will also be mapped, as little is known about how individual differences in hand and motor functions of the clinically used assessments with the brain outcome measures. Elucidating brain outcome measures that relate to developing motor functions is crucial for using early MRI scans in medical evaluations. Such patterns could help predict a child's motor skills and how these might develop, which could be important for directing future interventions.

METHODS

The following methods will be used for the NIBS-CP study:

Magnetic Resonance Imaging (MRI) The MRI protocol consists of several different structural MRI sequences, diffusion-weighted imaging, and MR-spectroscopy. Children will be scanned using a 3 Tesla MR scanner. The MRI protocol takes approximately 45 minutes. If the infant/toddler moves during a specific sequence, the specific sequence will be redone, if possible. In such cases, the protocol may take up to 1 hour. Earplugs as well as headphones will help minimize the scanner-related noise experienced by the infant/toddler.

Structural magnetic resonance imaging (sMRI) gives high-resolution images of the brain anatomy with different contrasts (e.g., T1-weighted and T2-weighted images). This kind of scanning allows for the quantification of different brain measures, such as volumes of specific brain regions and cortical thickness estimates. Moreover, sMRI provides the images that the neuroradiologist will read and use diagnostically.

Diffusion-weighted imaging (DWI) provides information about the microstructure of both gray and white matter tissue as well as structural connectivity.

Proton MR spectroscopy (MRS) will yield a metabolic profile of the basal ganglia/internal capsule region, including markers of neuronal integrity (e.g., N-acetyl-aspartate and glutamate), and glial markers (e.g., myoinositol). Voxels will include the left or right basal ganglia and internal capsule, to capture the metabolic profile in this region.

Sequences will be ordered so that the most important sequences (sMRI > DWI > MRS) will be acquired first, to optimize the chances of getting the sequences needed for diagnostic purposes for the infants at high risk of CP needing a diagnostic scan.

Neurological assessments Hammersmith Infant Neurological Examination (HINE) will be conducted by a pediatrician at Hvidovre Hospital for the typically developing infants and within the CP-EDIT study for the infants at risk for CP.

Motor and cognitive assessments

Motor and cognitive assessments of the typically developing infants will be conducted by physio- and occupational therapists at Hvidovre Hospital. Infants at risk for CP will undergo the same tests within the CP-EDIT protocol. The following motor and cognitive tests are included:

* Alberta Infant Motor Scale (AIMS)
* Hand Assessments for Infants (HAI)
* Bayley Scales of Infant and Toddler Development, 4th Edition (BSID-4)
* Peabody Developmental Motor Scales, 2nd Edition (PDMS-2)

Questionnaires

Neuropsychological data will be collected using the following parent-reported questionnaires for all participants (typically developing and at-risk for CP):

* Ages & Stages (ASQ). There are two questionnaires, one assessing motor and cognitive development and one assessing socio-emotional development.
* Demographics & Background

STUDY OUTLINE

Study outline for the typically developing infants in NIBS-CP:

The NIBS-CP study consists of three assessment rounds:

* Round 1 (inclusion) at age 3-6 months (infants may range from age 2 months or to 11 months), including MRI, HINE, AIMS, HAI, and Demographics & Background.
* Round 2 at age 12 months, including MRI, AIMS, HAI, ASQ, and Demographics & Background.
* Round 3 at age 24 months, including MRI, PDMS-2, ASQ, BSID-4, and Demographics & Background.

Study outline for CP-EDIT participants in NIBS-CP:

Families enrolled in CP-EDIT will be asked to participate in three MRI scans at age 2-11 months (Round 1, inclusion), age 12 months (Round 2, first follow-up), and age 24 months (Round 3, second follow-up) in parallel to CP-EDIT. Participation in NIBS-CP only includes MRI scans and parent-reported questionnaires (ASQ and Demographics & Background).

STATISTICAL CONSIDARATIONS Longitudinal data will be collected from 200 infants. Infant cohorts are typically smaller than adult cohorts, because of the challenges of MR-scanning this age group (Korom et al., 2022). The success rate of the scans is expected to be around 75% for sMRI, 60% for DWI, and 50% for MRS. The decline in success rate is due to the order of the sequences, given the higher risk of infants waking up the longer the scan time.

Statistical analyses will be conducted in statistical software tools, such as R and SPSS, and in image analysis specific tools, such as FreeSurfer and FSL. We will use e.g., analysis of covariance (ANCOVA) and multiple linear regression for cross-sectional data, and e.g., linear mixed models, generalized additive mixed models (GAMM), and repeated measurements analysis of variance (ANOVA) for longitudinal data

CP patient cohorts are biologically and clinically heterogeneous. Thus, in addition to examining differences in group averages, the normative modeling framework will be used (Rutherford et al., 2023, 2022) to quantify heterogeneity in structural brain measures by mapping structural brain changes at the level of the individual. Normative modeling is a leading tool in precision medicine, as it allows for elucidating differences at the individual level, mapped in relation to a reference model of normative data, similar to height growth charting in pediatric medicine. Here, normative modeling involves charting percentiles of variation across a population in terms of mappings of brain measures, or e.g., between brain measures and motor functioning. Publicly available datasets, such as the Healthy Brain and Child Development (HBCD) study, will be used to enhance our training dataset. In all models with MRI, age, sex, and variables estimating subject motion during MRI will be utilized as covariates.

ELIGIBILITY:
Inclusion Criteria High-Risk population:

Group: 'Newborn-detectable risk-pathway'

* Preterm birth with gestational age below 32 weeks
* Birth weight below 1500 g
* Moderate to severe brain injury (A label of moderate to severe brain injury was considered if there was Papile grade three to four intraventricular haemorrhage, cystic periventricular leukomalacia, neonatal stroke, term hypoxic-ischaemic encephalopathy (≥35 weeks gestation at birth) or other significant neurological condition)
* History (e.g., neonatal seizures, ECMO, meningitis, kernicterus, severe hypoglycemia) or neurological risk factors (malformations in CNS, increased tone)

Group: 'Infant detectable risk-pathway'

* Inability to sit independently by age 9 months
* Hand function asymmetry or crawl asymmetry
* Inability to take weight through the plantar surface of the feet
* History (e.g., as above) or neurological risk factors

Additional inclusion criteria for inclusion in NIBS-CP for both CP-risk groups:

- Consent to health-relevant information on clinical findings being passed on to the medical doctors in CP-EDIT and/or their primary care physician.

Inclusion Criteria Typically developing infant population:

* Born >37 weeks
* Uneventful birth
* No known history of brain injury
* No neurological condition
* Consent to health-relevant information on clinical findings being passed on to their primary care physician or relevant medical doctors, e.g., neuropaediatrician.

Exclusion Criteria (all groups):

* Infants have any MRI contraindications, e.g., pacemaker or other implanted electronic devices.
* Families do not speak or understand Danish.
* Families do not wish to be informed about incidental findings on the MRI, or scores within the clinical range in the neurological, motor, or cognitive assessments.

Ages: 2 Months to 11 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Infants at risk of cerebral palsy:
  160 infants with a high risk of CP will be enrolled in CP-EDIT (ClinicalTrials.gov ID NCT05835674). At least 2/3 are expected to be from the 'new-born detectable risk pathway' and less than 1/3 from the 'infant-detectable pathway'. At inclusion, infants will mainly be 3-6 months of age, though the age range between 2-11 months is accepted. It is expected that at least 50-60 of the high-risk infants will participate in the NIBS-CP study, with an upper limit of 100 infants.
  Typically developing infants:
  To establish a Danish normative sample of early brain development and a control group to the CP-EDIT cohort, approx. 140-150 typically developing infants will be recruited to NIBS-CP (approx. 200 infants when combining the high-risk and typically developing groups). The age range and mean age of the typically developing infants will be matched to that of the high-risk infants.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-06-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Diffusion-weighted magnetic resonance imaging | Baseline, 12 months, 24 months
  Microstructural measures obtained from fixel-based and tensor-based analysis.
Brain volumetric measures | Baseline, 12 months, 24 months
  Total brain volume, cortex volume, and white matter volume, as well as regional grey matter volume of cortical parcels and subcortical grey matter structures measured in mm3
Cortical thickness | Baseline, 12 months, 24 months
  Global and regional measures of apparent cortical thickness measured in mm
Brain connectivity measures | Baseline, 12 months, 24 months
  Brain connectivity measures obtained from structural covariance and tractography-based connectivity analyses
Indices of myelination | Baseline, 12 months, 24 months
  T1/T2 contrast in grey and white matter regions
MR-spectroscopy measures | Baseline, 12 months, 24 months
  Brain metabolic measures (metabolites: NAA, choline, creatine, myoinositol, lactate) obtained from voxels containing the basal ganglia and thalamus in the left and right hemispheres.
Surface area | Baseline, 12 months, 24 months
  Global and regional surface area measured in mm2

SECONDARY OUTCOMES:
Hand assessment for infants (HAI) | Baseline, 12 months
  The HAI measures the degree and quality of goal-directed actions performed with each hand separately as well as with both hands together. The HAI is scored on 17 items (12 unimanual and 5 bimanual)
Alberta Infant Motor Scale (AIMS) | Baseline, 12 months
  The AIMS is an observational assessment scale that measures gross motor maturation in infants from birth through independent walking. The scale consists of 58 items organized into four positions: prone, supine, sitting, and standing. Each item describes three aspects of motor performance - weight-bearing, posture, and antigravity movements.
Peabody Developmental Motor Scales (PDMS-2) | 24 months
  PDMS-2 is an in-depth assessment of gross and fine motor skills of children from birth through 5 years.
Bayley Scales of Infant and Toddler Development, Fourth Edition (BSID-4) | 24 months
  BSID-4 is a standardized and norm-referenced assessment that measures the cognitive, motor, language, and social-emotional development of infants and toddlers aged 0-3 years.
Ages & Stages (ASQ) | 12 months, 24 months
  ASQ is a parent-rated questionnaire for screening young children's developmental milestones between the ages of 1 month to 5½ years. There are two main questionnaires, one assessing motor and cognitive development and one assessing socio-emotional development.
Hammersmith Infant Neurological Examination (HINE) | Baseline, 24 months
  HINE is a standardized and scorable neurological examination used in the diagnosis of CP up to the age of 24 months. The HINE detects CP with more than 90% accuracy and provides objective information about severity.

CONTACTS AND LOCATIONS:
Overall Officials: Kathrine Skak Madsen, PhD, Principal Investigator — Senior Researcher
Locations (1):
- Danish Research Centre for Magnetic Resonance, Hvidovre, Capital Region, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wagenaar N, Verhage CH, de Vries LS, van Gasselt BPL, Koopman C, Leemans A, Groenendaal F, Benders MJNL, van der Aa NE. Early prediction of unilateral cerebral palsy in infants at risk: MRI versus the hand assessment for infants. Pediatr Res. 2020 Apr;87(5):932-939. doi: 10.1038/s41390-019-0664-5. Epub 2019 Nov 13. PMID 31722367
- [Background] Korom M, Camacho MC, Filippi CA, Licandro R, Moore LA, Dufford A, Zollei L, Graham AM, Spann M, Howell B; FIT'NG; Shultz S, Scheinost D. Dear reviewers: Responses to common reviewer critiques about infant neuroimaging studies. Dev Cogn Neurosci. 2022 Feb;53:101055. doi: 10.1016/j.dcn.2021.101055. Epub 2021 Dec 27. PMID 34974250
- [Background] Rutherford S, Barkema P, Tso IF, Sripada C, Beckmann CF, Ruhe HG, Marquand AF. Evidence for embracing normative modeling. Elife. 2023 Mar 13;12:e85082. doi: 10.7554/eLife.85082. PMID 36912775
- [Background] Rutherford S, Kia SM, Wolfers T, Fraza C, Zabihi M, Dinga R, Berthet P, Worker A, Verdi S, Ruhe HG, Beckmann CF, Marquand AF. The normative modeling framework for computational psychiatry. Nat Protoc. 2022 Jul;17(7):1711-1734. doi: 10.1038/s41596-022-00696-5. Epub 2022 Jun 1. PMID 35650452